CLINICAL TRIAL: NCT06312566
Title: A Multiple-Dose, Open-Label, Randomized, 2-Way Cross-Over Study to Assess the Bioequivalence Between Brivaracetam Tablet and Dry Syrup in Healthy Male Japanese Participants
Brief Title: A Study to Assess the Bioequivalence Between Brivaracetam Tablet and Dry Syrup in Healthy Japanese Male Study Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EP0231
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Healthy Study Participants
Keywords: brivaracetam; Healthy Study Participants; Phase 1; BRV
MeSH Terms: interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A-B (Experimental): Study participants randomized to this arm will receive multiple doses of brivaracetam tablet (Treatment A) as reference and multiple doses of brivaracetam dry syrup (Treatment B) as test in the treatment sequence A-B at pre-specified timepoints.
  Interventions: Drug: brivaracetam (BRV) tablet; Drug: brivaracetam (BRV) dry syrup
- Treatment B-A (Experimental): Study participants randomized to this arm will receive multiple doses of brivaracetam tablet (Treatment A) as reference and multiple doses of brivaracetam dry syrup (Treatment B) as test in the treatment sequence B-A at pre-specified timepoints.
  Interventions: Drug: brivaracetam (BRV) tablet; Drug: brivaracetam (BRV) dry syrup

INTERVENTIONS:
Drug: brivaracetam (BRV) tablet — Study participants will receive multiple-doses of brivaracetam tablet (reference - Treatment A) administered orally.
  Other Names: BRV; Briviact
Drug: brivaracetam (BRV) dry syrup — Study participants will receive multiple-doses of brivaracetam dry syrup (test - Treatment B) administered orally.
  Other Names: BRV

SUMMARY:
The purpose of the study is to demonstrate the bioequivalence between the BRV tablet and BRV dry syrup after multiple oral doses in healthy male Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be between 20 to 50 years of age (inclusive) at the time of signing the informed consent form (ICF)
* Participant is of Japanese descent as evidenced by appearance and verbal confirmation of familial heritage (ie, participant has all 4 Japanese grandparents born in Japan)
* Participant is male

Exclusion Criteria:

* Participant has a known hypersensitivity to any components of the investigational medicinal product (IMP) formulations
* Participant has participated in another study of an IMP (and/or an investigational device) within the previous 30 days or within 5 times the half-life (whichever is longer) of the first dose of BRV in this study or is currently participating in another study of an IMP (and/or an investigational device)
* Participant tests positive for alcohol and/or prohibited concomitant drugs (including cotinine) at the Screening Visit or on Day-1
* Participant has donated blood or plasma or has experienced blood loss ≥400 mL within 90 days, ≥200 mL within 30 days, or has donated any blood or plasma within 14 days before first administration of IMP
* Participant is a current smoker or has used nicotine-containing products (eg, tobacco, patches, gum) within 30 days before the first administration of IMP

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- EP0231 1, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in March 2024 and concluded in June 2024.
Pre-assignment Details: The Participant Flow refers to the Randomized Set.
Groups:
- Sequence Brivaracetam (BRV) Tablet - BRV Dry Syrup: Dosing period 1 consisted of 5 days (Day -1 [1 day before administration of IMP] to Day 4): On Day 1 and Day 2 each participant received a dose of BRV 50 mg tablet formulation twice daily; on Day 3, each participant received a single morning dose of BRV 50 mg tablet formulation. Dosing period 2 consisted of 5 days (Day -1 [1 day before administration of IMP] to Day 4): On Day 1 and Day 2 each participant received a dose of BRV 50mg as dry syrup twice daily; on Day 3, each participant received a single morning dose of BRV 50 mg as dry syrup. The final IMP administration in Dosing Period 1 and the first investigational medicinal product (IMP) administration in Dosing Period 2 were separated by a washout period of 6-10 days.
- Sequence BRV Dry Syrup - BRV Tablet: Dosing period 1 consisted of 5 days (Day -1 [1 day before administration of IMP] to Day 4): on Day 1 and Day 2 each participant received a dose of BRV 50 mg as dry syrup twice daily. On Day 3, each participant received a single morning dose of BRV 50 mg as dry syrup. Dosing period 2 consisted of 5 days (Day -1 [1 day before administration of IMP] to Day 4): On Day 1 and Day 2 each participant received a dose of BRV 50 mg tablet formulation twice daily; on Day 3 of Dosing Period 2, each participant received a single morning dose of BRV 50 mg tablet formulation. The final IMP administration in Dosing Period 1 and the first IMP administration in Dosing Period 2 were separated by a washout period of 6-10 days.
Period: Overall Study
Arm/Group | Sequence Brivaracetam (BRV) Tablet - BRV Dry Syrup | Sequence BRV Dry Syrup - BRV Tablet
Started | 32 | 32 (1 participant randomized to the BRV dry syrup - BRV tablet treatment sequence and discontinued the study due to a protocol violation before BRV tablet administration in Dosing Period 2.)
Completed | 32 | 31
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refers to the safety set (SS) which included all randomized participants who received at least 1 dose of the investigational medicinal product (IMP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence Brivaracetam (BRV) Tablet - BRV Dry Syrup | Sequence BRV Dry Syrup - BRV Tablet | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (9.8) | 33.8 (9.1) | 33.6 (9.4)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  19 - 65 years | 32 | 32 | 64
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 32 | 32 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 32 | 32 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration at Steady State [Cmax(ss)] After Multiple Doses of Brivaracetam
Description: Cmax,ss is the maximum plasma concentration of brivaracetam at steady state.
Time Frame: Day 1: before the morning and evening doses (0 and 12 hr); Day 2: before the morning and evening doses (24 and 36 hr); Day 3: Predose (48 hr) and 10 min, 15 min, 20 min, 30 min, 45 min, 60 min, 75 min, 90 min, 2 hr, 6 hr, 9 hr, and 12 hr postdose
Population: Pharmacokinetic (PK) set included all participants who were randomized, received at least 1 dose of active IMP, and had at least 1 quantifiable post-baseline PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Groups:
- BRV Tablet: Participants received BRV 50 mg tablet twice daily on Day 1 and Day 2 followed by a single administration on Day 3, under fasting conditions in Dosing Period 1 and Dosing Period 2 of the study.
- BRV Dry Syrup: Participants received BRV 50 mg dry syrup twice daily on Day 1 and Day 2 followed by a single administration on Day 3, under fasting conditions in Dosing Period 1 and Dosing Period 2 of the study.
Arm/Group | BRV Tablet | BRV Dry Syrup
Number analyzed (Participants) | 63 | 64
microgram per milliliter (μg/mL) | 2.963 (24.1) | 2.878 (19.5)
Statistical Analysis 1: Comparison: BRV Tablet vs BRV Dry Syrup; Test type: Equivalence — Bioequivalence between the BRV tablet (reference) and BRV dry syrup (test) formulations were concluded if the 92.016% CI limits for Cmax,ss was within the 0.80 to 1.25 range; Linear mixed model analysis; Ratio of Dry Syrup/ Tablet = 0.9726, 92.016% CI 2-sided [0.9257 to 1.022]

2. Primary Outcome: Area Under the Curve During a Dosing Interval at Steady State [AUC(Tau)] After Multiple Doses of Brivaracetam
Description: AUCtau was area under the curve during a dosing interval at steady state of brivaracetam.
Time Frame: as for outcome 1
Population: PK set included all participants who were randomized, received at least 1 dose of active IMP, and had at least 1 quantifiable post-Baseline PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*μg/mL
Arm/Group | BRV Tablet | BRV Dry Syrup
Number analyzed (Participants) | 63 | 64
hours*μg/mL | 18.55 (17.4) | 18.53 (16.8)
Statistical Analysis 1: Comparison: BRV Tablet vs BRV Dry Syrup; Test type: Equivalence — Bioequivalence between the BRV tablet (reference) and BRV dry syrup (test) formulations were concluded if the 90% CI limits for AUC(tau) was within the 0.80 to 1.25 range; Ratio of Dry Syrup/ Tablet = 0.9999, 92.016% CI 2-sided [0.9881 to 1.012]

3. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP. A TEAE was defined as any AE with a start date/time on or after the first dose of IMP or any unresolved event already present before administration of IMP that worsens in intensity following exposure to IMP.
Time Frame: From Baseline to end of Safety Follow-up (up to 25 days)
Population: SS included all randomized participants who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | BRV Tablet | BRV Dry Syrup
Number analyzed (Participants) | 63 | 64
percentage of participants | 4.8 | 10.9

4. Secondary Outcome: Percentage of Study Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: A TEAE was defined as any AE with a start date/time on or after the first dose of IMP or any unresolved event already present before administration of IMP that worsens in intensity following exposure to IMP. A serious adverse event (SAE) was defined as any untoward medical occurrence that at any dose:
  Results in death, Is life-threatening, Requires in patient hospitalization or prolongation of existing hospitalization, Is a congenital anomaly or birth defect, Results in persistent disability/incapacity Is an infection that requires treatment parenteral antibiotics, Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline to end of Safety Follow-up (up to 25 days)
Population: SS included all randomized participants who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | BRV Tablet | BRV Dry Syrup
Number analyzed (Participants) | 63 | 64
percentage of participants | 0 | 0

5. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Discontinuation
Description: Percentage of participants with TEAEs leading to discontinuation were reported.
Time Frame: From Baseline to end of Safety Follow-up (up to 25 days)
Population: SS included all randomized participants who received at least 1 dose of the IMP.
Measure: Number; unit: percentage of participants
Arm/Group | BRV Tablet | BRV Dry Syrup
Number analyzed (Participants) | 63 | 64
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline to end of Safety Follow-Up (up to 25 days)
Description: A TEAE was defined as any AE with a start date/time on or after the first dose of IMP or any unresolved event already present before administration of IMP that worsened in intensity following exposure to IMP. SS included all randomized participants who received at least 1 dose of the IMP.
Arm/Group | BRV Tablet | BRV Dry Syrup
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/64
Other Adverse Events (participants affected / at risk) | 2/63 | 6/64
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRV Tablet (N=63) | BRV Dry Syrup (N=64)
Dizziness (Nervous system disorders) | 2 (3) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT06312566/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT06312566/SAP_001.pdf